CLINICAL TRIAL: NCT04963049
Title: Effects of Exercising With a Facemask on Cardiorespiratory Performance at Intensities Below and Above the Ventilatory Threshold
Brief Title: Effects of Facemask on Cardiorespiratory Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, João Pedro Jesus, Principal Investigator, Faculdade de Motricidade Humana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23/2021
Record Dates: First submitted 2021-06-28; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Facemask Impact on Cardiorespiratory Performance
MeSH Terms: interventions — Clinical Protocols; Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- With Mask (Experimental)
  Interventions: Other: Protocol with Mask

INTERVENTIONS:
Other: Protocol with Mask — Look at differences in group with facemask and no mask

SUMMARY:
The purpose of the study is to explore whether using a surgical facemask impacts performance in response exercise below vs. above the ventilatory threshold (VT). The investigatores also aim to explore the impact of sexual dimorphism in the physiological response to exercise performed within these specific intensities. Finally, the onvestigators intend to examine whether the effects of wearing a facemask affect physiological recovery at cessation of exercise

DETAILED DESCRIPTION:
Tests will be carried out during the afternoon period (between 13.00 and 16.00 h), in a laboratory with an environmental temperature between 22 and 24 ºC and a relative humidity between 44 and 56%.

Each participant will be tested on 3 non-consecutive days. On the first day, a Graded Exercise Testin (GXT) will be performed, to measure VO2max and to enable the individualization of intensities according to the VT of each participant. (Silva et al., 2011). Then, in a randomized (computer generated algorithm) counterbalanced manner, all participants performed resting and standardized cycle-ergometer submaximal protocols on two different conditions (with and without facemask), within a 1-week period. On the first visit, body mass measurements will be taken, to the nearest 0.01 kg, on a digital scale (BG 42, Breuer GmbH, Söflinger, Germany) with the participants wearing light-weight clothes and no shoes. Measurements of standing height will be limited to the first visit and taken to the nearest 0.5 cm using a stadiometer. Body Mass index (BMI) will be calculated by dividing the participants' mass in kilograms by the square of their height in meters. Then, after a brief warm-up period, each participant will perform a maximal cycle-ergometer test consisting of a ramp protocol to volitional exhaustion.

One of our purposes is to determine the impact of exercising with a facemask on physiological recovery. For this reason, measurements, within each submaximal testing session (with and without a facemask), will be taken using a standardized timeline designed to allow measuring recovery postsubmaximal exercise and compare it with a resting baseline time point. Specifically, testing will begin with a 10-min resting period in the seated position (baseline). Subsequently, participants will exercise either without (control) or with (experimental) a surgical facemask at an intensity below the VT and recover for another 10 min. Then, each participant will exercise at an intensity above the VT until volitional exhaustion and this will be followed by 10 min of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18 to 30 years old adults

Exclusion Criteria:

* Potential participants, with body mass index (BMI) > 24.9 kg.m2 will be excluded. Additional exclusionary criteria will include active smoking status, known metabolic disease, cardiovascular disease, respiratory disorders including asthma; and any orthopedic issues that would limit exercise performance.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Differences in VO2max | 1 week
  Differences between the two groups in the vo2max and
Differences in Heart Rate | 1 week
  Differences between the two groups in the Heart Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade Motricidade Humana, Oeiras, Cruz Quebrada, Portugal

REFERENCES:
- [Derived] Jesus JP, Gomes M, Dias-Goncalves A, Correia JM, Pezarat-Correia P, Mendonca GV. Effects of surgical masks on the responses to constant work-rate cycling performed at different intensity domains. Clin Physiol Funct Imaging. 2022 Jan;42(1):43-52. doi: 10.1111/cpf.12734. Epub 2021 Nov 20. PMID 34753208